CLINICAL TRIAL: NCT02334007
Title: Extended Low-Molecular Weight Heparin VTE Prophylaxis in the Thoracic Surgery Population, a Prospective, Randomized Controlled Study
Brief Title: Extended Low-Molecular Weight Heparin VTE Prophylaxis in Thoracic Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SJHH_VTEpro001
Record Dates: First submitted 2014-12-18; First posted 2015-01-08 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Venous Thromboembolism; Lung Neoplasms; Pulmonary Embolism
Keywords: venous thromboembolism prophylaxis; deep vein thrombosis; pulmonary embolism; lung resection; low molecular weight heparin
MeSH Terms: conditions — Venous Thromboembolism; Lung Neoplasms; Pulmonary Embolism; Venous Thrombosis | interventions — Dalteparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LMWH: Dalteparin (Experimental): Consenting patients undergoing lung resection will receive standard postoperative thromboprophylaxis in hospital until the time of discharge. Subsequently, patients will be administered LMWH for duration of 30 days as outpatients.
  Interventions: Drug: LMWH: Dalteparin
- Placebo (Placebo Comparator): After undergoing lung resection these patients will research standard post-op TE prophylaxis and upon discharge will be administered a placebo injection of subcutaneous saline for 30 days duration.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: LMWH: Dalteparin — Dalteparin is a low-molecular weight heparin. The dosage used will be 5000 units once daily (administered as a subcutaneous injection). This is an established prophylactic dose used to prevent the incidence of VTE after surgery.
  Other Names: Fragmin
  Arms: LMWH: Dalteparin
Other: Placebo — Upon hospital discharge, half of the patients will be assigned to receive saline placebo injections for up to 35 days after surgery. These injections will have no effect.
  Arms: Placebo

SUMMARY:
After any surgery, there is a risk of venous thromboembolism (VTE), including Deep Vein Thrombosis (DVT) in the major veins of the legs and Pulmonary Embolus (PE) in the lungs. These clots are usually prevented by the administration of low-molecular-weight heparin, a blood thinner that prevents clotting. In most surgical specialties like thoracic or vascular surgery, this treatment is used until patients are discharged from the hospital. However, in orthopaedic surgery, there is strong evidence that longer term preventative treatment up to 35 days after hospital discharge helps to reduce VTE occurrences. In thoracic surgery, there is an even greater risk of developing PE because of the surgical stress, the common presence of cancer and direct damage to blood vessels in the lung during surgery. Despite the potential utility, the use of extended VTE prevention has never been evaluated in the thoracic surgery population. If extended treatment prevents clots, more patients will avoid complications related to VTE. There is currently very limited information available on the incidence of venous thromboembolism (VTE) in patients undergoing lung cancer resection and the utility of extended thromboprophylaxis (ET) in this patient population. Furthermore, in contrast to patients undergoing orthopaedic surgery where ET has become standard of care, duration of thromboprophylaxis is not well defined in this patient population. Therefore, there is a clear need to systematically evaluate the effects of extended VTE prophylaxis on the incidence of VTE in the post-op population.

DETAILED DESCRIPTION:
There is currently very limited information available on the incidence of venous thromboembolism (VTE) in patients undergoing lung cancer resection and the utility of extended thromboprophylaxis (ET) in this patient population. Furthermore, in contrast to patients undergoing orthopaedic surgery where ET has become standard of care, duration of thromboprophylaxis is not well defined in this patient population. Therefore, there is a clear need to systematically evaluate the effects of extended VTE prophylaxis on the incidence of VTE in the post-op population.

As a pilot study, the primary outcome will involve feasibility measures. The investigators aim to measure the proportion of recruitment within each centre, compliance, loss to follow-up, and tolerability of the intervention, defined as the number and severity of per-defined adverse events. The primary outcome of interest for the future full-scale trial is the 30-day incidence rate of VTE following extended 30-day prophylaxis (defined as pulmonary emboli or deep venous thromboembolism of the lower limb as detected by CT (Computed Tomography) pulmonary angiography and full leg Doppler ultrasound, respectively) following lung resection for malignancies.

The proposed pilot project is a multicenter blinded placebo-controlled randomized controlled pilot clinical trial assessing the feasibility and effectiveness of extended-duration VTE prophylaxis (30 days post-operatively) vs. short-term prophylaxis restricted to in-hospital stay with outpatient injected placebo, in patients undergoing lung resection for lung cancer or metastatic disease. All patients will receive both a peri-operative dose followed by postoperative VTE prophylaxis for the duration of their hospital stay. Those who were randomized to prolonged prophylaxis will continue the same dosage regime for an overall of 30 days, whereas the control group will receive placebo injections for the same duration of time.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be at least 18 years of age.
2. Patient may be of either gender.
3. Patients must be diagnosed with resectable lung cancer or metastatic lung disease eligible to complete metastasectomy.
4. Patients must be undergoing one of the following surgeries: segmentectomy, wedge resection, lobectomy, bilobectomy or pneumonectomy.
5. Patients must be competent to understand consent documents.

Exclusion Criteria:

1. All patients with known allergic or anaphylactic reaction to contrast dye, heparin or low molecular weight heparin (LMWH).
2. Patients must not be under current anticoagulation for venous thromboembolism or other medical conditions.
3. Patients must not have known renal impairment (defined as estimated glomerular filtration rate of less than 30ml/min/m2 as calculated by the Cockcroft-Gault method) either pre-operatively or as identified based on blood work obtained prior to the scheduled 30-day post-operative scan.
4. Patients must not have known hepatic failure, with international normalized ratio (INR) of >1.5.
5. Patients with history of, or ongoing liver disease, manifested as ascites or previous peritoneal tapping for ascites.
6. Patients must not be pregnant or planning to become pregnant.
7. Patients must not have been diagnosed or treated for VTE in the past 3 months prior to surgery.
8. Patients must not have a known, objectively confirmed bleeding disorder.
9. Patients must not have a present or previous increase risk of haemorrhage.
10. Patients must not have a history of previous heparin induced thrombocytopenia.
11. Baseline platelet count <75,000 but transient, recovered thrombocytopenia associated with chemotherapy will not be a basis for exclusion.
12. Patients must not have previously inserted inferior vena cava filter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-09; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Composite primary outcome: To determine the feasibility of a full scale trial by determining the recruitment rates and loss to follow up rates | 1-1.5 years
  Measuring accrual rates, patient compliance, adherence to protocol, any-cause loss to follow up, tolerability of the intervention (safety), adverse events, and coordination of participating centre infrastructure

SECONDARY OUTCOMES:
Clinical outcome:Comparison of Incidence of DVT and PE at 30 days after surgery between control and interventional arms (Outcome will be measured by a Chest Computed Tomography (CT) scan with PE contrast protocol and a full leg doppler ultrasound) | 30 days, +/- 5 days
  As a pilot study, there is an insufficient number of patients to definitively calculate incidence and compare treatment arms. However, this is a key outcome and the study will seek to determine this outcome. Outcome will be measured by a Chest Computed Tomography (CT) scan with PE contrast protocol and a full leg doppler ultrasound at approximately 30 days after surgery to seek the occurrence of clots
Occurrence of major and minor bleeding at 30 days post-surgery, +/- 5 days | 30 days after surgery
  Bleeding is a potential adverse event of Fragmin use. Major bleeding is defined as: Fatal bleeding OR Critical bleeding in a symptomatic area (intracranial, intraspinal, retroperitoneal, pericardial, or intramuscular with compartment syndrome) OR Bleeding causing a fall in hemoglobin level of 2g/dL or more as measured by a blood test at 30 days follow up, OR Bleeding requiring a blood transfusion of at least 2 units of packed red blood cells (excluding transfusions administered intra-operatively or 6-hrs post-operatively since these could not be impacted by post-surgical prophylaxis). Minor bleeding is defined as any bleeding episode not classified as major.
Comparison of mortality within 90 days of surgery between control and interventional arms | 90 days
  Both procedure-specific and all-cause mortality rates will be calculated
Number of cases of heparin administration related HIT (Heparin Induced Thrombocytopenia) within 90 days of surgery | 90 days
Number of participants with study-related adverse events within 90 days of surgery | 90 days
Comparison of non-DVT-associated PE events (those occurring without an antecedent DVT) between control and interventional arms | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Shargall, MD, FRCSC, FCCP, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Toronto General Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fahim C, Hylton D, Simunovic M, Agzarian J, Finley C, Hanna WC, Shargall Y. Development of the IRIS-AR strategy: an intervention to improve rates of accrual and retention for the VTE-PRO randomized controlled trial. Trials. 2019 Jul 19;20(1):447. doi: 10.1186/s13063-019-3536-8. PMID 31324209